CLINICAL TRIAL: NCT05401734
Title: Robot Assisted Gait Training in Persons With a Spinal Cord Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Thomas More Kempen (Other)
Collaborators: AZ Herentals (Unknown)
Responsible Party: Principal Investigator, Lieven De Maesschalck, Principal investigator / Innovationmanager, Thomas More Kempen
Other Study IDs: S58158
Record Dates: First submitted 2022-05-18; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: SCI - Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Cohort 1: Approximately 10 persons with a SCI will be included in the study. All participants are persons included in the RAGT program organized by the To Walk Again Postrehabilitation Centre. The recruitment will be performed by word of mouth. Participants utilizing the Eksoskeleton at the To Walk Again Postrehabilitation Centre will be asked if they are willing to participate in this study. Participation will be strictly voluntary
  Interventions: Device: Observation and follow up measurement
- Cohort 2: Approximately 10 persons with a SCI will be included in the study. All participants are persons included in the RAGT program organized by the To Walk Again Postrehabilitation Centre. The recruitment will be performed by word of mouth. Participants utilizing the Eksoskeleton at the To Walk Again Postrehabilitation Centre will be asked if they are willing to participate in this study. Participation will be strictly voluntary
  Interventions: Device: Observation and follow up measurement
- Cohort 3: Approximately 10 persons with a SCI will be included in the study. All participants are persons included in the RAGT program organized by the To Walk Again Postrehabilitation Centre. The recruitment will be performed by word of mouth. Participants utilizing the Eksoskeleton at the To Walk Again Postrehabilitation Centre will be asked if they are willing to participate in this study. Participation will be strictly voluntary
  Interventions: Device: Observation and follow up measurement

INTERVENTIONS:
Device: Observation and follow up measurement — The measured variables include:
  Questionnaires
  * Health related quality of life (Health Related Quality of Life Questionnaire)
  * Physical activity level (Physical Activity Scale for Persons with Impairments and Disabilities)
  * Walking ability (Walking Index for Spinal Cord Injury)
  * Independence in activities of daily living (SCIM III Questionnaire)
  * Pain (International SCI Pain Basic Data Set)
  * Resilience (Resilience Scale)
  * Bowel and bladder function (Neurogenic Bowel Dysfunction score, International Consultation on Incontinence Modular Questionnaire - Lower Urinary Tract Symptoms)
  Measurements:
  * Muscular strength and joint ROM (Manual Muscle Testing)
  * Spasticity (Modified Ashworth Scale)
  * Walking parameters (walking time, crutch position, forward and lateral center of gravity shift, step length and height, swing phase, walking speed)
  * Cardiovascular response (blood pressure, heart frequency, blood lactate concentration and Borg RPE score)

SUMMARY:
Over the past decade, RAGT has emerged as a promising method for improving ambulation after spinal cord injury (SCI). Early reports of this therapy were very promising, yet a recent study suggested that even though RAGT may improve locomotor ability in the acute SCI population, it appears less functional to more conventional forms of ambulation such as wheelchair propulsion.

What most of these studies have neglected to address, however, is the efficacy of RAGT as a therapeutic exercise intervention for the SCI population. Indeed, persons with SCI lead by definition a sedentary lifestyle. This reduced activity can lead to a variety of secondary health complications, including an increased risk for cardiovascular disease, spasticity, altered muscle composition and reduced joint range of motion (ROM), increased risk for pressure sores, reduced bone mineral density, increased risk for osteoporosis, and bladder and bowel dysfunction. In addition, psychological components such as body image, self-esteem, self-efficacy, psychological well-being and quality of life in general may be affected.

Consequently, before RAGT is dismissed as an expensive but perhaps not superior alternative to conventional rehabilitation strategies after SCI, the potential effect of this therapy on a variety of health-related outcomes needs to be considered, and the potential physiological and psychological benefits associated with this whole-body upright exercise therapy may justify its use in both the acute and chronic SCI populations. Several investigations have already indicated that regular exposure to RAGT results in some very significant health-related benefits that may decrease the aforementioned risk of secondary health complications. To our knowledge however, longitudinal effect studies in the SCI population have not yet been conducted, and further studies are needed to provide definitive evidence. It can be assumed that such insights may further optimize long-term health benefits, but also the cost-benefit ratio of RAGT. In addition, a detailed analysis of RAGT parameters (walking time, crutch position, forward and lateral center of gravity shift, step length and height, swing phase, walking speed, etc.) and the direct cardiovascular response (heart frequency, blood pressure, blood lactate concentration) to RAGT have not yet been conducted.

The purpose of this research project is therefore to investigate the longitudinal effect of RAGT on the psychological well-being (Quality of Life, pain, fatigue), independence in activities of daily living, muscular strength and joint range of motion (ROM), and bladder and bowel function in persons with SCI.

DETAILED DESCRIPTION:
Over the past decade, RAGT has emerged as a promising method for improving ambulation after spinal cord injury (SCI). Early reports of this therapy were very promising, yet a recent study suggested that even though RAGT may improve locomotor ability in the acute SCI population, it appears less functional to more conventional forms of ambulation such as wheelchair propulsion.

What most of these studies have neglected to address, however, is the efficacy of RAGT as a therapeutic exercise intervention for the SCI population. Indeed, persons with SCI lead by definition a sedentary lifestyle. This reduced activity can lead to a variety of secondary health complications, including an increased risk for cardiovascular disease, spasticity, altered muscle composition and reduced joint range of motion (ROM), increased risk for pressure sores, reduced bone mineral density, increased risk for osteoporosis, and bladder and bowel dysfunction. In addition, psychological components such as body image, self-esteem, self-efficacy, psychological well-being and quality of life in general may be affected.

Consequently, before RAGT is dismissed as an expensive but perhaps not superior alternative to conventional rehabilitation strategies after SCI, the potential effect of this therapy on a variety of health-related outcomes needs to be considered, and the potential physiological and psychological benefits associated with this whole-body upright exercise therapy may justify its use in both the acute and chronic SCI populations. Several investigations have already indicated that regular exposure to RAGT results in some very significant health-related benefits that may decrease the aforementioned risk of secondary health complications. To our knowledge however, longitudinal effect studies in the SCI population have not yet been conducted, and further studies are needed to provide definitive evidence. It can be assumed that such insights may further optimize long-term health benefits, but also the cost-benefit ratio of RAGT. In addition, a detailed analysis of RAGT parameters (walking time, crutch position, forward and lateral center of gravity shift, step length and height, swing phase, walking speed, etc.) and the direct cardiovascular response (heart frequency, blood pressure, blood lactate concentration) to RAGT have not yet been conducted.

The purpose of this research project is therefore to investigate the longitudinal effect of RAGT on the psychological well-being (Quality of Life, pain, fatigue), independence in activities of daily living, muscular strength and joint range of motion (ROM), and bladder and bowel function in persons with SCI over a period of 2 years in several cohorts. We will measure every three months. Patients will be asked to fill in the questionnaires 3, 6 9, 12, 15, 18, 21 and 24 months after inclusion. Additionally the patients will we asked to fill in his medication intake in the follow-up system.

ELIGIBILITY:
Inclusion Criteria:

* SCI
* Bone density

Exclusion Criteria:

* osteoporosis
* length more than 2 meter

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Approximately 50 persons with a SCI will be included in the study. All participants are persons included in the RAGT program organized by the To Walk Again Postrehabilitation Centre. The recruitment will be performed by word of mouth. Participants utilizing the Eksoskeleton at the To Walk Again Postrehabilitation Centre will be asked if they are willing to participate in this study. Participation will be strictly voluntary
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2012-02-01; Primary Completion 2014-10-30 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
ROM (Range of Motion) | 3 months
  Range of Motion. We measure the range of motion of the legs with a Goniometer every three months. Our goal is to see if there is an improvement due to the robot asssited gait training
ROM (Range of Motion) | 6 months
  Range of Motion. We measure the range of motion of the legs with a Goniometer every three months. Our goal is to see if there is an improvement due to the robot asssited gait training
ROM (Range of Motion) | 9 months
  Range of Motion. We measure the range of motion of the legs with a Goniometer every three months. Our goal is to see if there is an improvement due to the robot asssited gait training
ROM (Range of Motion) | 12 months
  Range of Motion. We measure the range of motion of the legs with a Goniometer every three months. Our goal is to see if there is an improvement due to the robot asssited gait training
ROM (Range of Motion) | 15 months
  Range of Motion. We measure the range of motion of the legs with a Goniometer every three months. Our goal is to see if there is an improvement due to the robot asssited gait training
ROM (Range of Motion) | 18 months
  Range of Motion. We measure the range of motion of the legs with a Goniometer every three months. Our goal is to see if there is an improvement due to the robot asssited gait training
ROM (Range of Motion) | 21 months
  Range of Motion. We measure the range of motion of the legs with a Goniometer every three months. Our goal is to see if there is an improvement due to the robot asssited gait training
ROM (Range of Motion) | 24 months
  Range of Motion. We measure the range of motion of the legs with a Goniometer every three months. Our goal is to see if there is an improvement due to the robot asssited gait training
WHOQOL | 3 months
  World Health Organization Qualitiy of Life Questionnaire - BREF (WHOQoL-BREF). We are using the WHOQOL-Bref instrument (questionnaire). The WHOQOL is a quality of life assessment developed by the WHOQOL Group with fifteen international field centres, simultaneously, in an attempt to develop a quality of life assessment that would be applicable cross-culturally. WHOQOL-BREF is a generic health related QoL measure consisting of 26 items divided into 6 sub-scales. It has 4 domains namely physical health, psychological health, social relationship and environment, and 2 individual subscales on overall quality of life and general health. It can be self-administered and has good internal consistency (0.75-0.87). The higher the score, the more QOL. Each item is scored between 1 and 5. This scores will be translated to a score between 0-100 based on the manual for the general score and each subdomain score. This questionnaire will be filled in every three months by the patient.
WHOQOL | 6 months
  World Health Organization Qualitiy of Life Questionnaire - BREF (WHOQoL-BREF). We are using the WHOQOL-Bref instrument (questionnaire). The WHOQOL is a quality of life assessment developed by the WHOQOL Group with fifteen international field centres, simultaneously, in an attempt to develop a quality of life assessment that would be applicable cross-culturally. WHOQOL-BREF is a generic health related QoL measure consisting of 26 items divided into 6 sub-scales. It has 4 domains namely physical health, psychological health, social relationship and environment, and 2 individual subscales on overall quality of life and general health. It can be self-administered and has good internal consistency (0.75-0.87). The higher the score, the more QOL. Each item is scored between 1 and 5. This scores will be translated to a score between 0-100 based on the manual for the general score and each subdomain score. This questionnaire will be filled in every three months by the patient.
WHOQOL | 9 months
  World Health Organization Qualitiy of Life Questionnaire - BREF (WHOQoL-BREF). We are using the WHOQOL-Bref instrument (questionnaire). The WHOQOL is a quality of life assessment developed by the WHOQOL Group with fifteen international field centres, simultaneously, in an attempt to develop a quality of life assessment that would be applicable cross-culturally. WHOQOL-BREF is a generic health related QoL measure consisting of 26 items divided into 6 sub-scales. It has 4 domains namely physical health, psychological health, social relationship and environment, and 2 individual subscales on overall quality of life and general health. It can be self-administered and has good internal consistency (0.75-0.87). The higher the score, the more QOL. Each item is scored between 1 and 5. This scores will be translated to a score between 0-100 based on the manual for the general score and each subdomain score. This questionnaire will be filled in every three months by the patient.
WHOQOL | 12 months
  World Health Organization Qualitiy of Life Questionnaire - BREF (WHOQoL-BREF). We are using the WHOQOL-Bref instrument (questionnaire). The WHOQOL is a quality of life assessment developed by the WHOQOL Group with fifteen international field centres, simultaneously, in an attempt to develop a quality of life assessment that would be applicable cross-culturally. WHOQOL-BREF is a generic health related QoL measure consisting of 26 items divided into 6 sub-scales. It has 4 domains namely physical health, psychological health, social relationship and environment, and 2 individual subscales on overall quality of life and general health. It can be self-administered and has good internal consistency (0.75-0.87). The higher the score, the more QOL. Each item is scored between 1 and 5. This scores will be translated to a score between 0-100 based on the manual for the general score and each subdomain score. This questionnaire will be filled in every three months by the patient.
WHOQOL | 15 months
  World Health Organization Qualitiy of Life Questionnaire - BREF (WHOQoL-BREF). We are using the WHOQOL-Bref instrument (questionnaire). The WHOQOL is a quality of life assessment developed by the WHOQOL Group with fifteen international field centres, simultaneously, in an attempt to develop a quality of life assessment that would be applicable cross-culturally. WHOQOL-BREF is a generic health related QoL measure consisting of 26 items divided into 6 sub-scales. It has 4 domains namely physical health, psychological health, social relationship and environment, and 2 individual subscales on overall quality of life and general health. It can be self-administered and has good internal consistency (0.75-0.87). The higher the score, the more QOL. Each item is scored between 1 and 5. This scores will be translated to a score between 0-100 based on the manual for the general score and each subdomain score. This questionnaire will be filled in every three months by the patient.
WHOQOL | 18 months
  World Health Organization Qualitiy of Life Questionnaire - BREF (WHOQoL-BREF). We are using the WHOQOL-Bref instrument (questionnaire). The WHOQOL is a quality of life assessment developed by the WHOQOL Group with fifteen international field centres, simultaneously, in an attempt to develop a quality of life assessment that would be applicable cross-culturally. WHOQOL-BREF is a generic health related QoL measure consisting of 26 items divided into 6 sub-scales. It has 4 domains namely physical health, psychological health, social relationship and environment, and 2 individual subscales on overall quality of life and general health. It can be self-administered and has good internal consistency (0.75-0.87). The higher the score, the more QOL. Each item is scored between 0 and 5. This scores will be translated to a score between 0-100 based on the manual for the general score and each subdomain score. This questionnaire will be filled in every three months by the patient.
WHOQOL | 21 months
  World Health Organization Qualitiy of Life Questionnaire - BREF (WHOQoL-BREF). We are using the WHOQOL-Bref instrument (questionnaire). The WHOQOL is a quality of life assessment developed by the WHOQOL Group with fifteen international field centres, simultaneously, in an attempt to develop a quality of life assessment that would be applicable cross-culturally. WHOQOL-BREF is a generic health related QoL measure consisting of 26 items divided into 6 sub-scales. It has 4 domains namely physical health, psychological health, social relationship and environment, and 2 individual subscales on overall quality of life and general health. It can be self-administered and has good internal consistency (0.75-0.87). The higher the score, the more QOL. Each item is scored between 1 and 5. This scores will be translated to a score between 0-100 based on the manual for the general score and each subdomain score. This questionnaire will be filled in every three months by the patient.
WHOQOL | 24 months
  World Health Organization Qualitiy of Life Questionnaire - BREF (WHOQoL-BREF). We are using the WHOQOL-Bref instrument (questionnaire). The WHOQOL is a quality of life assessment developed by the WHOQOL Group with fifteen international field centres, simultaneously, in an attempt to develop a quality of life assessment that would be applicable cross-culturally. WHOQOL-BREF is a generic health related QoL measure consisting of 26 items divided into 6 sub-scales. It has 4 domains namely physical health, psychological health, social relationship and environment, and 2 individual subscales on overall quality of life and general health. It can be self-administered and has good internal consistency (0.75-0.87). The higher the score, the more QOL. Each item is scored between 1 and 5. This scores will be translated to a score between 0-100 based on the manual for the general score and each subdomain score. This questionnaire will be filled in every three months by the patient.
IPA | 3 months
  Participation of daily life (IPA). This is a valid and reliable questionnaire (Impact on participation and autonomy). This questionnaire is based on the international classification of human functioning. The goal of of this questionnaire is to have a clear image on the way your healthy status influences your abilities to live your life and how you experience this feeling. This questionnaire consist of 32 items divided in 5 domains. (Autonomy outside, family roll, autonomy inside, social relations, work and education). Scores for each item are between 0 to 4. The lower the score the better; the higher the score the more barriers. For each domain a mean score between 0 and 4 will be calculated.
IPA | 6 months
  Participation of daily life (IPA). This is a valid and reliable questionnaire (Impact on participation and autonomy). This questionnaire is based on the international classification of human functioning. The goal of of this questionnaire is to have a clear image on the way your healthy status influences your abilities to live your life and how you experience this feeling. This questionnaire consist of 32 items divided in 5 domains. (Autonomy outside, family roll, autonomy inside, social relations, work and education). Scores for each item are between 0 to 4. The lower the score the better; the higher the score the more barriers. For each domain a mean score between 0 and 4 will be calculated.
IPA | 9 months
  Participation of daily life (IPA). This is a valid and reliable questionnaire (Impact on participation and autonomy). This questionnaire is based on the international classification of human functioning. The goal of of this questionnaire is to have a clear image on the way your healthy status influences your abilities to live your life and how you experience this feeling. This questionnaire consist of 32 items divided in 5 domains. (Autonomy outside, family roll, autonomy inside, social relations, work and education). Scores for each item are between 0 to 4. The lower the score the better; the higher the score the more barriers. For each domain a mean score between 0 and 4 will be calculated.
IPA | 12 months
  Participation of daily life (IPA). This is a valid and reliable questionnaire (Impact on participation and autonomy). This questionnaire is based on the international classification of human functioning. The goal of of this questionnaire is to have a clear image on the way your healthy status influences your abilities to live your life and how you experience this feeling. This questionnaire consist of 32 items divided in 5 domains. (Autonomy outside, family roll, autonomy inside, social relations, work and education). Scores for each item are between 0 to 4. The lower the score the better; the higher the score the more barriers. For each domain a mean score between 0 and 4 will be calculated.
IPA | 15 months
  Participation of daily life (IPA). This is a valid and reliable questionnaire (Impact on participation and autonomy). This questionnaire is based on the international classification of human functioning. The goal of of this questionnaire is to have a clear image on the way your healthy status influences your abilities to live your life and how you experience this feeling. This questionnaire consist of 32 items divided in 5 domains. (Autonomy outside, family roll, autonomy inside, social relations, work and education). Scores for each item are between 0 to 4. The lower the score the better; the higher the score the more barriers. For each domain a mean score between 0 and 4 will be calculated.
IPA | 18 months
  Participation of daily life (IPA). This is a valid and reliable questionnaire (Impact on participation and autonomy). This questionnaire is based on the international classification of human functioning. The goal of of this questionnaire is to have a clear image on the way your healthy status influences your abilities to live your life and how you experience this feeling. This questionnaire consist of 32 items divided in 5 domains. (Autonomy outside, family roll, autonomy inside, social relations, work and education). Scores for each item are between 0 to 4. The lower the score the better; the higher the score the more barriers. For each domain a mean score between 0 and 4 will be calculated.
IPA | 21 months
  Participation of daily life (IPA). This is a valid and reliable questionnaire (Impact on participation and autonomy). This questionnaire is based on the international classification of human functioning. The goal of of this questionnaire is to have a clear image on the way your healthy status influences your abilities to live your life and how you experience this feeling. This questionnaire consist of 32 items divided in 5 domains. (Autonomy outside, family roll, autonomy inside, social relations, work and education). Scores for each item are between 0 to 4. The lower the score the better; the higher the score the more barriers. For each domain a mean score between 0 and 4 will be calculated.
IPA | 24 months
  Participation of daily life (IPA). This is a valid and reliable questionnaire (Impact on participation and autonomy). This questionnaire is based on the international classification of human functioning. The goal of of this questionnaire is to have a clear image on the way your healthy status influences your abilities to live your life and how you experience this feeling. This questionnaire consist of 32 items divided in 5 domains. (Autonomy outside, family roll, autonomy inside, social relations, work and education). Scores for each item are between 0 to 4. The lower the score the better; the higher the score the more barriers. For each domain a mean score between 0 and 4 will be calculated.
Bowel and bladder function | 3 months
  We will use the Neurogenic Bowel Dysfunction score. This valid and reliable questionnaire consist of 10 items. The minimum score is 0 the maximum score is 47. The higher the score, the more discomfort. 0-6: very less; Score 7-9: Minimal; Score 10-13: Moderate, Score 14+: severe. For urinary we use the International Consultation on Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life Module (ICIQ-LUTSqol). The ICIQ-LUTSqol is a psychometrically robust patient-completed questionnaire evaluating quality of life (QoL) in urinary incontinent patients. The ICIQ-LUTSqol is the King's Health Questionnaire (KHQ) adapted for use within the ICIQ structure and provides a measure to assess the impact of urinary incontinence on quality of life with particular reference to social effects. It consists 20 items sore between 0-10). 19-76 overall score with greater values indicating increased impact on quality of life.
Bowel and bladder function | 6 months
  We will use the Neurogenic Bowel Dysfunction score. This valid and reliable questionnaire consist of 10 items. The minimum score is 0 the maximum score is 47. The higher the score, the more discomfort. 0-6: very less; Score 7-9: Minimal; Score 10-13: Moderate, Score 14+: severe. For urinary we use the International Consultation on Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life Module (ICIQ-LUTSqol). The ICIQ-LUTSqol is a psychometrically robust patient-completed questionnaire evaluating quality of life (QoL) in urinary incontinent patients. The ICIQ-LUTSqol is the King's Health Questionnaire (KHQ) adapted for use within the ICIQ structure and provides a measure to assess the impact of urinary incontinence on quality of life with particular reference to social effects. It consists 20 items sore between 0-10). 19-76 overall score with greater values indicating increased impact on quality of life.
Bowel and bladder function | 9 months
  We will use the Neurogenic Bowel Dysfunction score. This valid and reliable questionnaire consist of 10 items. The minimum score is 0 the maximum score is 47. The higher the score, the more discomfort. 0-6: very less; Score 7-9: Minimal; Score 10-13: Moderate, Score 14+: severe. For urinary we use the International Consultation on Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life Module (ICIQ-LUTSqol). The ICIQ-LUTSqol is a psychometrically robust patient-completed questionnaire evaluating quality of life (QoL) in urinary incontinent patients. The ICIQ-LUTSqol is the King's Health Questionnaire (KHQ) adapted for use within the ICIQ structure and provides a measure to assess the impact of urinary incontinence on quality of life with particular reference to social effects. It consists 20 items sore between 0-10). 19-76 overall score with greater values indicating increased impact on quality of life.
Bowel and bladder function | 12 months
  We will use the Neurogenic Bowel Dysfunction score. This valid and reliable questionnaire consist of 10 items. The minimum score is 0 the maximum score is 47. The higher the score, the more discomfort. 0-6: very less; Score 7-9: Minimal; Score 10-13: Moderate, Score 14+: severe. For urinary we use the International Consultation on Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life Module (ICIQ-LUTSqol). The ICIQ-LUTSqol is a psychometrically robust patient-completed questionnaire evaluating quality of life (QoL) in urinary incontinent patients. The ICIQ-LUTSqol is the King's Health Questionnaire (KHQ) adapted for use within the ICIQ structure and provides a measure to assess the impact of urinary incontinence on quality of life with particular reference to social effects. It consists 20 items sore between 0-10). 19-76 overall score with greater values indicating increased impact on quality of life.
Bowel and bladder function | 15 months
  We will use the Neurogenic Bowel Dysfunction score. This valid and reliable questionnaire consist of 10 items. The minimum score is 0 the maximum score is 47. The higher the score, the more discomfort. 0-6: very less; Score 7-9: Minimal; Score 10-13: Moderate, Score 14+: severe. For urinary we use the International Consultation on Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life Module (ICIQ-LUTSqol). The ICIQ-LUTSqol is a psychometrically robust patient-completed questionnaire evaluating quality of life (QoL) in urinary incontinent patients. The ICIQ-LUTSqol is the King's Health Questionnaire (KHQ) adapted for use within the ICIQ structure and provides a measure to assess the impact of urinary incontinence on quality of life with particular reference to social effects. It consists 20 items sore between 0-10). 19-76 overall score with greater values indicating increased impact on quality of life.
Bowel and bladder function | 18 months
  We will use the Neurogenic Bowel Dysfunction score. This valid and reliable questionnaire consist of 10 items. The minimum score is 0 the maximum score is 47. The higher the score, the more discomfort. 0-6: very less; Score 7-9: Minimal; Score 10-13: Moderate, Score 14+: severe. For urinary we use the International Consultation on Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life Module (ICIQ-LUTSqol). The ICIQ-LUTSqol is a psychometrically robust patient-completed questionnaire evaluating quality of life (QoL) in urinary incontinent patients. The ICIQ-LUTSqol is the King's Health Questionnaire (KHQ) adapted for use within the ICIQ structure and provides a measure to assess the impact of urinary incontinence on quality of life with particular reference to social effects. It consists 20 items sore between 0-10). 19-76 overall score with greater values indicating increased impact on quality of life.
Bowel and bladder function | 21 months
  We will use the Neurogenic Bowel Dysfunction score. This valid and reliable questionnaire consist of 10 items. The minimum score is 0 the maximum score is 47. The higher the score, the more discomfort. 0-6: very less; Score 7-9: Minimal; Score 10-13: Moderate, Score 14+: severe. For urinary we use the International Consultation on Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life Module (ICIQ-LUTSqol). The ICIQ-LUTSqol is a psychometrically robust patient-completed questionnaire evaluating quality of life (QoL) in urinary incontinent patients. The ICIQ-LUTSqol is the King's Health Questionnaire (KHQ) adapted for use within the ICIQ structure and provides a measure to assess the impact of urinary incontinence on quality of life with particular reference to social effects. It consists 20 items sore between 0-10). 19-76 overall score with greater values indicating increased impact on quality of life.
Bowel and bladder function | 24 months
  We will use the Neurogenic Bowel Dysfunction score. This valid and reliable questionnaire consist of 10 items. The minimum score is 0 the maximum score is 47. The higher the score, the more discomfort. 0-6: very less; Score 7-9: Minimal; Score 10-13: Moderate, Score 14+: severe. For urinary we use the International Consultation on Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life Module (ICIQ-LUTSqol). The ICIQ-LUTSqol is a psychometrically robust patient-completed questionnaire evaluating quality of life (QoL) in urinary incontinent patients. The ICIQ-LUTSqol is the King's Health Questionnaire (KHQ) adapted for use within the ICIQ structure and provides a measure to assess the impact of urinary incontinence on quality of life with particular reference to social effects. It consists 20 items sore between 0-10). 19-76 overall score with greater values indicating increased impact on quality of life.

SECONDARY OUTCOMES:
Medication | 3 months
  Use of medication. We ask the patient to fill in an digital diary concerning medication intake. We ask digital information in a format with: Name of the medication, number of intake, prescription or not, regular or extra, reason.
Medication | 6 months
  Use of medication. We ask the patient to fill in an digital diary concerning medication intake. We ask digital information in a format with: Name of the medication, number of intake, prescription or not, regular or extra, reason.
Medication | 9 months
  Use of medication. We ask the patient to fill in an digital diary concerning medication intake. We ask digital information in a format with: Name of the medication, number of intake, prescription or not, regular or extra, reason.
Medication | 12 months
  use of medication. We ask the patient to fill in an diary concerning medication.
Medication | 15 months
  Use of medication. We ask the patient to fill in an digital diary concerning medication intake. We ask digital information in a format with: Name of the medication, number of intake, prescription or not, regular or extra, reason.
Medication | 18 months
  Use of medication. We ask the patient to fill in an digital diary concerning medication intake. We ask digital information in a format with: Name of the medication, number of intake, prescription or not, regular or extra, reason.
Medication | 21 months
  Use of medication. We ask the patient to fill in an digital diary concerning medication intake. We ask digital information in a format with: Name of the medication, number of intake, prescription or not, regular or extra, reason.
Medication | 24 months
  Use of medication. We ask the patient to fill in an digital diary concerning medication intake. We ask digital information in a format with: Name of the medication, number of intake, prescription or not, regular or extra, reason.

CONTACTS AND LOCATIONS:
Locations (1):
- De Maesschalck Lieven, Geel, Antwerp, Belgium